CLINICAL TRIAL: NCT00945243
Title: Prospective, Multi-Center Clinical Outcomes Study Evaluating the Zero-P PEEK for Anterior Cervical Interbody Fusion in the Treatment of Cervical Degenerative Disc Disease
Brief Title: Clinical Outcomes Study Evaluating the Zero-P PEEK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated early due to lower than expected enrollment rates.
Sponsor: Synthes USA HQ, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZeroP-021109
Record Dates: First submitted 2009-07-22; First posted 2009-07-24 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-09

CONDITIONS: Cervical Disc Disease
Keywords: SCDD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Other): Treatment of cervical DDD with the Zero-P device
  Interventions: Device: Zero-P

INTERVENTIONS:
Device: Zero-P — The Zero-P PEEK is a stand-alone device intended for use in cervical interbody fusion. The device consists of a plate and a spacer with four rigid screws to provide similar stability to a traditional cervical plate and interbody spacer. It is intended for use in skeletally mature patients with symptomatic cervical disc disease (SCDD) with accompanying radicular symptoms, at one level from C3 to C7.
  Other Names: Zero-P PEEK Spacer

SUMMARY:
This is a multi-center, prospective, outcomes study. In this study, the Zero-P PEEK implant will be used in patients undergoing ACDF for treatment of SCDD at a single level between C3 and C7. The cohort will be followed over time to twenty-four (24) months after surgery. Up to fifteen (15) sites will participate in this study. This is not a controlled study.

DETAILED DESCRIPTION:
This was a post-market study

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic cervical disc disease (SCDD) in only one vertebral level between C3-C7 requiring:

   1. Neck or arm (radicular) pain and/or
   2. Functional/neurological deficit confirmed by imaging (CT, MRI, X-Ray) of at least one of the following:

   i. herniated nucleus pulposus

   ii. spondylosis (defined by presence of osteophytes)

   iii. loss of disc height
2. NDI score greater than or equal to 15/50 (30%) (considered moderate disability);
3. Skeletally mature adult between the ages of 18-70 years at the time of surgery;
4. Has completed at least six (6) weeks of conservative therapy;
5. Psychosocially, mentally and physically able to fully comply with this protocol including adhering to scheduled visits, treatment plan, completing forms, and other study procedures;
6. Personally signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the study.

Exclusion Criteria:

1. More than one vertebral level to be fused;
2. Posterior instrumentation necessary at same level;
3. Has had previous surgery at the index level;
4. Has a fused level adjacent to the index level;
5. Active systemic or local infection;
6. Known or documented history of communicable disease, including AIDS or HIV;
7. Active hepatitis (receiving medical treatment within two years);
8. Active rheumatoid arthritis, non-controlled diabetes mellitus, or any other medical condition(s) that would represent a significant increase in surgical risk or interfere with normal healing;
9. Immunologically suppressed, or has received systemic steroids, excluding nasal steroids, at any dose daily for > 1 month within last 12 months;
10. Known history of Paget's disease, osteomalacia, or any other metabolic bone disease;
11. Osteopenia or Osteoporosis: A screening questionnaire for osteoporosis, SCORE (Simple Calculated Osteoporosis Risk Estimation), will be used to screen patients who require a DEXA bone mineral density measurement. If DEXA is required, exclusion will be defined as a DEXA bone density measured T score ≤ -1.0.
12. Previous known allergy to the materials contained in the device, such as polyetheretherketone (PEEK) or titanium alloy (TAN);
13. Morbid obesity defined as a body mass index > 40 kg/m2 or weight more than 100 pounds over ideal body weight;
14. Active malignancy. A patient with a history of any invasive malignancy (except non-melanoma skin cancer), unless treated with curative intent and there has been no clinical signs or symptoms of the malignancy for more than 5 years;
15. Current or recent history (within last 2 years) of substance abuse (e.g., recreational drugs, narcotics, or alcohol);
16. Pregnant or planning to become pregnant during study period;
17. Involved in study of another investigational product that may affect outcome;
18. History of psychosocial disorders that could prevent accurate completion of self reporting assessment scales;
19. Patients who are incarcerated.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2011-12-01 (Actual); Study Completion 2011-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lotito, Study Director — DePuy Synthes Assoc. Director Clinical Research
Locations (14):
- United States (14):
  - Neurospine, South East Alabama Medical Center, Dothan, Alabama
  - Barrow Neurosurgical Institute, Phoenix, Arizona
  - Newport Orthopaedics, Hoag Hospital, Newport Beach, California
  - Lyerly Neurosurgery Group, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Indiana Spine Center, Lafayette, Indiana
  - The Boston Spine Group, Newton, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Sierra Neurosurgery Group, Reno, Nevada
  - Reno Orthopaedic Clinic, Reno, Nevada
  - VSAS Orthopaedics, Allentown, Pennsylvania
  - Charleston Neurosurgical Associates, Charleston, South Carolina
  - Neurosurgery Northwest, Tacoma, Washington
  - Milwaukee Spinal Specialists, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Treatment of cervical DDD with the Zero-P device ACDF: The Zero-P PEEK is a stand-alone device intended for use in cervical interbody fusion. The device consists of a plate and a spacer with four rigid screws to provide similar stability to a traditional cervical plate and interbody spacer. It is intended for use in skeletally mature patients with symptomatic cervical disc disease (SCDD) with accompanying radicular symptoms, at one level from C3 to C7.
Period: Overall Study
Arm/Group | Treatment
Started | 11 (Enrolled and Treated Per Protocol)
Completed | 8
Not Completed | 3
Not completed — Study Terminated: Subjects Dispositioned | 3

BASELINE CHARACTERISTICS:
Population: Number of subjects enrolled and treated per protocol
Arm/Group | Treatment
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Neck Disability Index Scores
Description: Percentage of subjects who experienced a maintenance or improvement according to measures of pain and/or function.
Time Frame: 24 months
Population: 8 subjects had data at 24 months
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment
Number analyzed (Participants) | 8
percentage of subjects | 87.5

2. Secondary Outcome: Improvement in the Neck and Arm Visual Analog Pain Scale (VAS)
Description: Percentage of subjects who experienced a maintenance of improvement in VAS neck pain intensity, neck pain frequency, arm pain intensity, and/or arm pain frequency.
Time Frame: 24 months
Population: 8 subjects had data at 24 months.
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment
Number analyzed (Participants) | 8
percentage of subjects | 75.0

3. Secondary Outcome: Implant Related Complications
Description: Percentage of subjects who had an implant related complication
Time Frame: 24 months
Population: 11 subjects were enrolled and treated on protocol and were thus considered for safety information
Measure: Number; unit: percentage of subjects
Arm/Group | Treatment
Number analyzed (Participants) | 11
percentage of subjects | 0

ADVERSE EVENTS:
Time Frame: From enrollment out to 24 months
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 3/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=11)
Pain and/or Weakness (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 1 (1)
Cold Symptoms (Immune system disorders) | 1 (1)
Adjacent Level Surgery (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less